CLINICAL TRIAL: NCT06129266
Title: Oral Care With Breast Milk in Preterm Newborns Fed by Tube:A Randomized Controlled Study
Brief Title: Oral Care With Breast Milk in Preterm Newborns Fed by Tube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, Ayse Cuvadar, Assistant Professor, Karabuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13/38
Record Dates: First submitted 2023-11-04; First posted 2023-11-13 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Breastmilk; Oral Care
Keywords: breastmilk; oral care; newborn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention (Oral care with breastmilk) group (Experimental): Newborns selected according to the randomization group will receive nursing care, including oral care and feeding, from the same person twice a day, at 09:00 in the morning and 15:00 in the afternoon. Breast milk (BM) will be used for oral care. At each treatment, two ml BM should be dropped onto sterile gauze to clean the cheeks, tongue and palate. Process steps; After hand hygiene is achieved, it will be done using disposable gloves.
  Interventions: Other: oral care with breastmilk
- Routine maintenance group (No Intervention): No intervention will be applied to the control group other than oral care with sterile distilled water, which is routine clinical practice.

INTERVENTIONS:
Other: oral care with breastmilk — No intervention will be applied to the control group other than oral care with sterile distilled water, which is routine clinical practice.
  Other Names: routine maintenance
  Arms: İntervention (Oral care with breastmilk) group

SUMMARY:
It was conducted to evaluate Oral Care with Breast Milk in Preterm Newborns Fed by Tube

DETAILED DESCRIPTION:
Newborns selected according to the randomization group will receive nursing care, including oral care and feeding, from the same person twice a day, at 09:00 in the morning and 15:00 in the afternoon. Breast milk (BM) will be used for oral care. At each treatment, two ml BM should be dropped onto sterile gauze to clean the cheeks, tongue and palate. Process steps; After hand hygiene is achieved, it will be done using disposable gloves.

ELIGIBILITY:
Inclusion Criteria:

* -Staying in the neonatal intensive care unit
* Being fed by gavage
* Babies with no oral intake (nonperoral-NPO)
* Babies fed with breast milk and/or formula

Exclusion Criteria:

* Babies who are exclusively breastfed
* Cleft palate/lip
* Major congenital anomaly
* Intubated babies

Ages: 28 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Oral Care with Breast Milk in Tube-Fed Preterm Newborns: Randomized Controlled Study | from the same person twice a day, at 09:00 in the morning and 15:00 in the afternoon.
  Oral care

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)